CLINICAL TRIAL: NCT03592290
Title: Hemodynamics Monitoring During Lower Body Negative Pressure (LBNP) Induced Controlled Hypovolemia
Acronym: LBPN
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000020057; 000 (Other: CTGTY)
Record Dates: First submitted 2018-06-13; First posted 2018-07-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hypovolemia; Hemodynamic Instability
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lower body negative pressure — We will be monitoring the changes in central and peripheral monitors/waveforms during gradual hypovolemia induced by lower body negative pressure in healthy volunteers.

SUMMARY:
To monitor the changes in central and peripheral monitors/waveforms during gradual hypovolemia induced by lower body negative pressure in healthy volunteers.

DETAILED DESCRIPTION:
The primary aim of this research is to identify the most robust site for monitoring hypovolemia as well as assess changes in peripheral waveforms monitored by the pulse oximeter collected from different sites (finger, ear, forehead, and nose), blood pressure, cerebral oximetry and peripheral venous pressure during gradual hypovolemia induced by lower body negative pressure (LBNP) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 20-45 with

Exclusion Criteria:

* Pregnant women
* Under 20 years of age
* Subjects with coronary artery disease, diabetes, epilepsy and hypertension

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers aged 20-45 with no history of heart disease, diabetes, or hypertension. Pregnant women will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Identify the most robust site for monitoring hypovolemia utilizing pulse oximeter waveforms. | 2 years
  Data will be summarized using mean (SD) for normally distributed data, median (interquartile range) for non-normal data.
  linear regression method will be used to model the changes of our dependent variable from baseline during blood loss.

SECONDARY OUTCOMES:
Examine the relationship between central hemodynamic changes (cardiac output) with changes in respiratory variability of PPG waveforms collected from different sites during hypovolemia and fluid resuscitation | 2 years
  Data will be summarized using mean (SD) for normally distributed data, median (interquartile range) for non-normal data.
  linear regression method will be used to model the changes of our dependent variable from baseline during blood loss.

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Alian, MD, Principal Investigator — Yale University
Locations (1):
- John B. Pierce Laboratory, New Haven, Connecticut, United States